CLINICAL TRIAL: NCT03087318
Title: Sport as a Treatment in Chronic Diseases and Healthcare Sustainability: Sport 4 Health
Brief Title: Sport as a Treatment in Chronic Diseases and Healthcare Sustainability
Acronym: S4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC17.047; 2017-A00467-46 (Other: IdRCB)
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Obstructive Sleep Apnea; Overweight and Obesity
Keywords: Obstructive sleep apnea (OSA); Overweight and moderate obesity; Sport prescription; Physical activity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Overweight; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective, open, proof of concept study in overweight or moderate obese OSA patients, comparing 3 different programs of sport "prescription": patient's referred to a rehabilitation medical center, to a private sport club or to a sport association.
Masking Description: open, proof of concept study in overweight or moderate obese OSA patients,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rehabilitation medical center (Experimental): Physical activity:
  * 3 sessions / week at least
  * at least during 30 minutes each session
  * at least at 50% of the maximal HR(heart rate) measured during the exercise stress testing (from the screening)
  * during 3 months.
  Interventions: Behavioral: Physical activity
- Private sport club (Experimental): Physical activity:
  * 3 sessions / week at least
  * at least during 30 minutes each session
  * at least at 50% of the maximal HR(heart rate) measured during the exercise stress testing (from the screening)
  * during 3 months.
  Interventions: Behavioral: Physical activity
- Sport association (Experimental): Physical activity:
  * 3 sessions / week at least
  * at least during 30 minutes each session
  * at least at 50% of the maximal HR(heart rate) measured during the exercise stress testing (from the screening)
  * during 3 months.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Physical activity:
  * 3 sessions / week at least
  * at least during 30 minutes each session
  * at least at 50% of the maximal heart rate measured during the exercise stress testing (from the screening)
  * during 3 months.
  Other Names: Programs of sport "prescription"

SUMMARY:
Obesity, associated with obstructive sleep apnea (OSA) is often involved in cardiovascular diseases. In our study, we want to promote sport practice to reduce that burden in the first place, and all associated diseases (e.g. cardiovascular diseases) consequently. The aim of this clinical trial is to determine which type of program, conducted in a digital environment associating a mobile application and individual coaching, better improves exercise habits over a 3-month period in overweight or moderate obese OSA patients.

DETAILED DESCRIPTION:
With automation equipment and the comfort, it has brought, less natural physical activities are required and people do not take the time to do some. Therefore, obesity, associated with obstructive sleep apnea (OSA) up to 60% of cases, has become a heavy burden on the society and the healthcare system, besides the fact that it often involves cardiovascular diseases. Assistance is urgently needed and the investigators want to promote sport practice to reduce that burden in the first place, and all associated diseases (e.g. cardiovascular diseases) consequently. In order to do that, the investigators will integrate sport in the patient pathway and support in his/her involvement. This last point means that a link between medical and sport specialists should be established, and this is missing today.

This study aims to reconcile the world of patients and the world of sport, by offering a trajectory and an organization that help patients to initiate physical activity.

The investigators plan to measure the physical activity of overweight or moderate obese, apneic patients in the different programs at the end of the 3-month period by physical activity objective parameters: number of steps/day.

The secondary objectives of this study are to:

* Evaluate the effect of the different programs of sport "prescription" on patient motivation, over a 3-month period by a motivational questionnaire.
* Analyze the cost effectiveness of the different programs of sport "prescription" over a 3-month period.
* Evaluate the effect of the different programs of sport "prescription" on weight and blood pressure (BP), assessed by home self-measurements each month, over a 3-month period and recorded in the application.

ELIGIBILITY:
Inclusion Criteria:

* 25 y ≤ age ≤ 70 y
* 27 < BMI < 32
* Weight < 120 kg
* Apneic patient (Apnea-hypopnea index > 15/h) treated or not by CPAP (continuous positive airway pressure )
* Be able to practice sport (according to a Cardiologist decision)
* Be able to use the personal health monitoring devices jointly to a personal Touch phone
* Consenting patient based around Grenoble France
* Be legally able to give consent
* Person affiliated to social security

Exclusion Criteria:

* Being unable to understand, follow objectives and methods due to cognition or language problems
* Pregnant women, feeding and parturient
* Physical activity score > 9, calculated by Baecke's questionnaire (Annex 1)
* Subject under administrative or judicial control, person who are protected under the act.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
The physical activity of overweight or moderate obese OSA patients in the different programs will be estimated by physical activity objective parameters: number of steps/day. | at the end of the 3-month period
  The physical activity of overweight or moderate obese OSA patients in the different programs during the 3-month period will be estimated by physical activity objective parameters: heart rate, physical activity type, motion cadence (number of steps/day), energy expenditure, and sleep stage (measured at the end, by an actigraph integrated in the watch).

SECONDARY OUTCOMES:
Evaluation of the effect of the different programs of sport "prescription" on patient motivation | over a 3-month period
  The evaluation of the effect of the different programs of sport "prescription" on patient motivation will be assessed by a motivational questionnaire.
Cost effectiveness analysis of the different programs of sport "prescription" | over a 3-month period.
  Monthly cost of the subscription in the sport association, private sport club and rehabilitation medical center will be collected.
Evaluation of the effect of the different programs of sport "prescription" on weight and blood pressure (BP) | each month, over 3 months
  Monthly self measurement of weight and BP at home, recorded in the application

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, MD, PhD, Principal Investigator — University Hospital of Grenoble, France
Locations (1):
- University Hospital, Grenoble, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andrade FM, Pedrosa RP. The role of physical exercise in obstructive sleep apnea. J Bras Pneumol. 2016 Nov-Dec;42(6):457-464. doi: 10.1590/S1806-37562016000000156. PMID 28117479
- [Result] Borjesson M, Urhausen A, Kouidi E, Dugmore D, Sharma S, Halle M, Heidbuchel H, Bjornstad HH, Gielen S, Mezzani A, Corrado D, Pelliccia A, Vanhees L. Cardiovascular evaluation of middle-aged/ senior individuals engaged in leisure-time sport activities: position stand from the sections of exercise physiology and sports cardiology of the European Association of Cardiovascular Prevention and Rehabilitation. Eur J Cardiovasc Prev Rehabil. 2011 Jun;18(3):446-58. doi: 10.1097/HJR.0b013e32833bo969. PMID 21450560